CLINICAL TRIAL: NCT00667810
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy And Safety Trial Of Bapineuzumab (Aab-001, Eln115727) In Subjects With Mild to Moderate Alzheimer Disease Who Are Apolipoprotein E 4 Non-carriers
Brief Title: Study Evaluating The Efficacy And Safety Of Bapineuzumab In Alzheimer Disease Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated on August 6, 2012, because 2 large Phase 3 studies showed no clinical benefit. This decision was not based on any new safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3133K1-3000; B2521001 (Other: Alias Study Number); 2007-005994-79 (EudraCT Number); NCT00909623 (obsolete NCT alias)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Alzheimer Disease
Keywords: antibody; immunotherapy
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bapineuzumab 0.5 mg/kg (Experimental)
  Interventions: Drug: bapineuzumab
- Bapineuzumab 1.0 mg/kg (Experimental)
  Interventions: Drug: bapineuzumab
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bapineuzumab — Bapineuzumab 0.5 mg/kg administered by IV infusion approximately every 13 weeks through week 65.
  Other Names: AAB-001
  Arms: Bapineuzumab 0.5 mg/kg
Drug: bapineuzumab — Bapineuzumab 1.0 mg/kg administered by IV infusion approximately every 13 weeks through week 65.
  Other Names: AAB-001
  Arms: Bapineuzumab 1.0 mg/kg
Drug: placebo — Placebo will be administered by IV infusion approximately every 13 weeks through week 65.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of multiple doses of bapineuzumab in patients with mild to moderate Alzheimer Disease. Patients will receive either bapineuzumab or placebo. Each patient's participation will last approximately 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer Disease (AD), with Mini Mental State Examination (MMSE) score of 16-26, and brain magnetic resonance imaging (MRI) consistent with the diagnosis of AD
* Concurrent use of cholinesterase inhibitor or memantine allowed, if stable
* Caregiver will participate and be able to attend clinic visits with patient

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Contraindication to undergo brain MRI [e.g., pacemaker, cerebrospinal fluid (CSF) shunt, or foreign metal objects in the body]
* Women of childbearing potential

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2008-06; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (340):
- United States (160):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Jeffrey S. Gitt, DO, PC, Phoenix, Arizona
  - The Compounding Center (IP Mixing Only), Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - ATP Clinical Research, Incorporated, Costa Mesa, California
  - Pharmacology Research Institute, Encino, California
  - Margolin Brain Institute, Fresno, California
  - Infusion Care Pharmacey, Laguna Hills, California
  - Senior Clinical Trials, Incorporated, Laguna Hills, California
  - Faculty Physicians and Surgeons of Loma Linda University School of Medicine, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Coordinated Clinical Research, San Diego, California
  - LabCorp, San Diego, California
  - Sharp and Children's MRI Center, LLC, San Diego, California
  - Sharp Infusion Therapy Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Associated Neurologists, PC, Boulder, Colorado
  - The Mile High Research Center, Denver, Colorado
  - Associated Neurologists, PC, Danbury, Connecticut
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - Bendheim Cancer Center, Greenwich, Connecticut
  - Center for Healthy Aging, Greenwich, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Norman S. Werdiger, MD, New Haven, Connecticut
  - Institutional Review Board / Ethics Committee, New Haven, Connecticut
  - Yale PET Center, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - JEM Research Institute LLC, Atlantis, Florida
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Bradenton Research Center, Incorporated, Bradenton, Florida
  - North Broward Medical Center, Deerfield Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neurologic Consultants, P.A., Fort Lauderdale, Florida
  - MD Clinical, Hallandale, Florida
  - Renstar Medical Research, Ocala, Florida
  - Advanced Imaging, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Roskamp Institute, Sarasota, Florida
  - South Bay Internal Medicine, Sun City, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - NeuroTrials Research, Incorporated, Atlanta, Georgia
  - Columbus Diagnostic Center (MRI), Columbus, Georgia
  - Medical Research and Health Education Foundation, Incorporated, Columbus, Georgia
  - Dekalb Neurology Associates, LLC/NeuroStudies.net, LLC, Decatur, Georgia
  - NeuroStudies.net, Decatur, Georgia
  - Neurostudies.net, Lawerenceville, Georgia
  - Neurostudies.net, Lawrenceville, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Methodist Center for Senior Health, Peoria, Illinois
  - Methodist Medical Center Research Department, Peoria, Illinois
  - Methodist Diagnostic Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Psychology Associates, Mishawaka, Indiana
  - KU - Wichita, Wichita, Kansas
  - Drug Shipment/ Storage, Wichitia, Kansas
  - Four Rivers Clinical Research, Incorporated, Paducah, Kentucky
  - Radio Pharmacy, Paducah, Kentucky
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Research Associates Inc, New Orleans, Louisiana
  - James Gary Booker, MD, APMC, Shreveport, Louisiana
  - Foers Medical Arts Pharmacy, Bethesda, Maryland
  - CBH Health, LLC, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Bringham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - General Clinical Research Center, Boston, Massachusetts
  - IDS Pharmacy, Boston, Massachusetts
  - ActivMed Practices and Research, Inc., Haverhill, Massachusetts
  - Neurocare, Incorporated, Newton, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Michigan State University, Lansing, Michigan
  - Marty's Pharmacy, Flowood, Mississippi
  - Precise Research Centers, Flowood, Mississippi
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - Spectrum Home Solutions, Great Falls, Montana
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - Memory Enhancement Center of New Jersey, Inc., Toms River, New Jersey
  - Northeast Radiology, Brewster, New York
  - Neurological Care of Central New York, Liverpool, New York
  - AD-CARE, University of Rochester Medical Center, Rochester, New York
  - University of Rochester/Strong Memorial Hospital, Rochester, New York
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Clinical Trials of America, Incorporated, Hickory, North Carolina
  - The Compounding Pharmacy, Hickory, North Carolina
  - Carolina Neuropsychological Services, Inc., Raleigh, North Carolina
  - Healthsouth Blue Ridge Surgery Center, Raleigh, North Carolina
  - Raleigh Neurology Associates, PA, Raleigh, North Carolina
  - Wake Radiology Associates, Raleigh, North Carolina
  - Ohio State University Imaging at Martha Morehouse, Columbus, Ohio
  - The Ohio State University Hospitals Clinic, Columbus, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Professional Corporation of Psychiatry, Oklahoma City, Oklahoma
  - Red River Medical Recearch Center, LLC, Oklahoma City, Oklahoma
  - Flourish Integrative Pharmacy, Oklahoma City, Oklahoma
  - Providence Brain Institute, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Abington Neurological Associates, Abington, Pennsylvania
  - Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Hospital of the University of Pennslyvania, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania (PET), Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Investigational New Drug Services, IDS Pharmacy, Philadelphia, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - UPENN Clinical and Translational Research Center (CTRC), Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Simpson's Pharmacy, Pawtucket, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina Hospitals and Clinics, Charleston, South Carolina
  - Medical University of South Carolina Investigational Drug Service, Charleston, South Carolina
  - Radiant Research, Incorporated, Greer, South Carolina
  - Medical University of South Carolina, North Charleston, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - Austin Infusion Centers, Austin, Texas
  - Senior Adults Specialty Research, Austin, Texas
  - Texas Neurology, P.A., Dallas, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Vista Infusions, San Antonio, Texas
  - Inventive Infusion Solutions, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Southwestern Vermont Healthcare, Bennington, Vermont
  - The Memory Clinic, Bennington, Vermont
  - University of Virginia Neurology, Charlottesville, Virginia
  - University of Virginia General Clinical Research Center, Charlottesville, Virginia
  - University of Viriginia Investigational Pharmacy, Charlottesville, Virginia
  - Pacific Medical Centers, Bothell, Washington
  - Pacific Medical Centers, Seattle, Washington
- Argentina (2):
  - Cemic University Hospital, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
- Australia (8):
  - Gosford Hospital, Gosford, New South Wales
  - Hornsby Kuringai Hospital, Hornsby, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - CDAMS Ballarat Base Hospital, Ballarat, Victoria
  - Heidelberg Repatriation Hospital/ Medical and Cognitive Research Unit, West Heidelberg, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - McCusker Alzheimer's Research Foundation Inc., Nedlands, Western Australia
  - Royal Adelaide Hospital, Adelaide SA
- Belgium (6):
  - ZNA Middelheim / Neurologie, Antwerp
  - Az. St. Jan Ruddershove 35, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - University Hospital Gathuisberg, Leuven
  - H.-Hartziekenhuis Roeselare-Menen, Roeselare
- Canada (9):
  - Centre for Memory and Aging, North York, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre de Recherche ADAPRA Inc., L'Ancienne-Lorette, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Recherche Clinique de Neurologie, Montreal, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Chile (2):
  - Psicomedica Research Group, Santiago, Chile
  - Especialidades Medicas L&S, Santiago
- Croatia (2):
  - Sestre milosrdnice Zagreb, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Finland (2):
  - Turku University Hospital, Turku, Finland
  - Ita-Suomen Yliopisto, Kuopio
- France (19):
  - CHRU Hôtel Dieu, Rennes, Cedex
  - CHU de Dijon, Dijon, France
  - CHU Hopital Nord, Amiens
  - Hôpital Neurologique, Bron
  - CHU de Caen, Caen
  - Hôpitaux Civils de Colmar, Colmar
  - Hôpital Roger Salengro, Lille
  - Hopital Sainte Marguerite, Marseille
  - Hôpital la Timone, Marseille
  - CHU Hôpital Gui de Chaulliac, Montpellier
  - CHU Nord - Hôpital Guillaume et René Laënnec, Nantes - Saint Herblain
  - Hôpital Cimiez, Nice
  - Groupe Hospitalier Broca-La Rochefoucauld, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - CHU La Milétrie, Poitiers
  - C.H.U de Reims, Reims
  - CHU - Hopital Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse
  - CHU Purpan - Hôpital Casselardit, Toulouse
- Germany (4):
  - Klinik fur Psychiatrie und Psychotherapie, Berlin, State of Berlin
  - St. Josef-Klinikum, Bochum
  - Ortenau Klinikum, Offenburg
  - Universitaet Regensburg, Regensburg
- Italy (12):
  - Universita Politecnica delle Marche, Ancona
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Unita' Operativa Complessa di Neurologia, Catania
  - CeSI (Centro di Scienze dell'invecchiamento) -, Chieti
  - Universita degli Studi di Firenze, Florence
  - Ospedale S. Raffaele, Milan
  - Fondazione IRCCS- Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera S. Gerardo di Monza Università di Milano Bicocca, Monza
  - Ospedale S. Gerardo, Monza
  - Clinica Neurologica, Roma
  - Unita' Operativa C - Riabilitazione Neurologica, Roma
  - Universita degli Studi di Siena, Siena
- Japan (35):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tokyo Metoropolitan Health and Med. Treatment Co. Ebara Hosp, Ōta-ku, Tokyo
  - Yachiyo Hospital, Aichi
  - Kashiwado Hospital, Chiba
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Nippon Medical School Chiba Hokusoh Hospital, Chiba
  - National Hospital Organization Kokura Medical Center, Fukuoka
  - Maebashi Red Cross Hospital, Gunma
  - Gunma University Hospital, Gunma
  - Shinozuka Hospital, Gunma
  - National Hospital Organization Hiroshima-nishi Medical Ctr., Hiroshima
  - Kobe University Hospital, Hyōgo
  - Nishi-Kobe Medical Center, Hyōgo
  - Kobe City Hospital Org Kobe City Medical Cente West Hp, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Nippon Medical School Musashikosugi Hospital, Kanagawa
  - Yokohama City University Medical Center, Kanagawa
  - Shonan Atsugi Hospital, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Minami-Kyoto Hospital, Kyoto
  - National Hospital Organization Maizuru Medical Center, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Nagano
  - National Hospital Organization Niigata National Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - Okayama University Hospital, Okayama
  - National Hospital Organization Minami-Okayama Medical Center, Okayama
  - Osaka City University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Kansai Medical University Takii Hospital, Osaka
  - National HP.Org.Shizuoka Inst.Epilepsy,Neurological Disorder, Shizuoka
  - Juntendo University Hospital, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - National Hospital Organization Tokyo National Hospital, Tokyo
- Mexico (2):
  - OCA Hospital, Monterrey, Nuevo León
  - Instituto Biomedico de Investigacion A.C, Aguascalientes
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Kennemer Gasthuis, Haarlem
  - Medisch Centrum Leeuwarden, Leeuwarden
- New Zealand (2):
  - The Memory Clinic, Auckland, NZ
  - Signet Research, Christchurch
- Poland (6):
  - Szpital Uniwersytecki w Krakowie,Oddzial Kliniczny Klinik Chorób Wewnetrznych, Krakow, Poland
  - NZOZ "NEURO-KARD" "ILKOWSKI I PARTNERZY" Spolka Partnerska Lekarzy, Poznan, Poland
  - NZOZ Dom Suer Ryder, Pallmed Sp. z o.o., Bydgoszcz
  - NZOZ "SYNAPSA", ul. Niska 5/1, Kielce
  - Oddzial Neurologiczny i Udarowy Szpital Wolski im. dr Anny Gostynskiej,, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Katedra i Klinika, Warsaw
- Portugal (3):
  - Hospital Fernando da Fonseca, Amadora, Amadora
  - Hospitais Da Universidade De Coimbra, Coimbra, Coimbra District
  - Hospital Santa Maria, Lisbon, Lisbon District
- Russia (6):
  - Interregional clinicodiagnostic center, Kazan'
  - Nizhny Novgorod regional clinical hospital n.a. N.A.Semashko, Nizhny Novgorod
  - Saint-Petersburg State institution of healthcare, City geriatric medico-social center, Saint Petersburg
  - Saint Petersburg Psychoneurological Research Institute n.a. V.M.Bekhterev, Saint Petersburg
  - Saint-Petersburg Psychoneurological Research Institute n.a. V.M.Bekhterev, Saint Petersburg
  - Chair of nervous system diseases, Saint Petersburg
- Serbia (3):
  - Klinicki centar Vojvodine, Novi Sad, Vojvodina
  - Klinicki centar Srbije, Belgrade
  - Clinical Centre Kragujevac, Kragujevac
- Slovakia (7):
  - 1. Neurologicka klinika, Bratislava
  - Psychiatricka ambulancia, Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - Neurologicka klinika, Martin
  - Psychiatricka nemocnica Michalovce, n.o., Michalovce
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - Neurologicke oddelenie FNsP Zilina, Žilina
- South Africa (5):
  - Boithuso Caregivers, Johannesburg, Gauteng
  - The Osteoporosis and Memory Centre, Johannesburg, Gauteng
  - Denmar Clinic, Pretoria, Gauteng
  - St Augustine's Medical Centre 2, Durban, KwaZulu-Natal
  - Panorama Psychiatry and Memory Clinic, Panorama, Western Cape
- South Korea (2):
  - Seoul National University Bundang Hospital, Department of Psychiatry, Seongnam-si, Gyeonggi-do
  - KonKuk University Hospital, Department of NeuroPsychiatry, Seoul
- Spain (17):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - CLONUS, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Clínica CIMA, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Mutua de Terrasa, Terrassa, Barcelona
  - Hospital Divino Valles, Burgos, Burgos
  - Hospital Virgen del Puerto, Plasencia, Caceres
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital de Cruces, Barakaldo
  - Fundació ACE Institut Catala de Neurociences Aplicades, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
- Sweden (4):
  - Skanes Universitetssjukhus, Neuropsykiatriska, Malmo
  - PET center, Uppsala
  - The clinic: Minnes- och geriatrikmottagningen, Uppsala
  - MRI Dept: ORKI, Uppsala
- Switzerland (4):
  - Memory Clinic Neuro-Psychologie Zentrum, Basel, Canton of Basel-City
  - Hopitaux Universitaires de Geneve, Les Acacias, Canton of Geneva
  - CHUV Lausanne, Lausanne, Canton of Vaud
  - Hopitaux Universitaires de Geneve, Thonex-Geneva
- United Kingdom (12):
  - Glasgow Memory Clinic, Glasgow, Glasgow
  - MAC UK Neuroscience Ltd, Blackpool, Lancashire
  - Kings College Hospital, London, London
  - MAC UK Neuroscience, Ltd., Bradford, West Yorkshire
  - Clinical Investigation and Research Unit (CIRU), Brighton
  - Dept. of Neurosciences Charing Cross Hospital, London
  - Newcastle General Hospital, Newcastle upon Tyne
  - Northampton General Hospital NHS Trust, Northampton
  - Llandough Hospital, Penarth
  - Royal Hallamshire Hospital, Sheffield
  - Grenoside Grange Hospital, Sheffield
  - Kingshill Research Centre, Swindon

REFERENCES:
- [Derived] Vandenberghe R, Rinne JO, Boada M, Katayama S, Scheltens P, Vellas B, Tuchman M, Gass A, Fiebach JB, Hill D, Lobello K, Li D, McRae T, Lucas P, Evans I, Booth K, Luscan G, Wyman BT, Hua L, Yang L, Brashear HR, Black RS; Bapineuzumab 3000 and 3001 Clinical Study Investigators. Bapineuzumab for mild to moderate Alzheimer's disease in two global, randomized, phase 3 trials. Alzheimers Res Ther. 2016 May 12;8(1):18. doi: 10.1186/s13195-016-0189-7. PMID 27176461
- [Derived] Lacey L, Bobula J, Rudell K, Alvir J, Leibman C. Quality of Life and Utility Measurement in a Large Clinical Trial Sample of Patients with Mild to Moderate Alzheimer's Disease: Determinants and Level of Changes Observed. Value Health. 2015 Jul;18(5):638-45. doi: 10.1016/j.jval.2015.03.1787. Epub 2015 Apr 10. PMID 26297092
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133K1-3000&StudyName=Study%20Evaluating%20The%20Efficacy%20And%20Safety%20Of%20Bapineuzumab%20In%20Alzheimer%20Disease%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated on 06 August 2012 due to lack of clinical efficacy observed in completed studies ELN115727-301 (ApoE4 non-carriers) and ELN115727-302. A total of 329 participants had completed the study up to and including Week 78 before the decision was taken to terminate the study.
Pre-assignment Details: The study originally included bapineuzumab 2.0 mg/kg dose level, which was discontinued on 02 April 2009 based on input from independent safety monitoring committee. It was estimated at the time that about 10 participants received 2.0mg/kg. These participants are not included in the efficacy analyses.
Groups:
- Bapineuzumab 0.5 mg/kg: Participants received 0.5 mg/kg bapineuzumab by intravenous (IV) infusion every 13 weeks, for a total of 6 infusions over the course of the study. A final follow-up visit was performed at Week 78, 13 weeks after the last infusion.
- Bapineuzumab 1.0 mg/kg: Participants received 1.0 mg/kg bapineuzumab by IV infusion every 13 weeks, for a total of 6 infusions over the course of the study. A final follow-up visit was performed at Week 78, 13 weeks after the last infusion.
- Placebo: Participants received placebo by IV infusion every 13 weeks, for a total of 6 infusions over the course of the study. A final follow-up visit was performed at Week 78, 13 weeks after the last infusion.
- Bapineuzumab 2.0 mg/kg: Participants received 2.0 mg/kg bapineuzumab by IV infusion every 13 weeks, for a total of 6 infusions over the course of the study. A final follow-up visit was performed at Week 78, 13 weeks after the last infusion.
Period: Overall Study
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo | Bapineuzumab 2.0 mg/kg
Started | 269 | 264 | 346 | 11
Treated | 267 | 263 | 344 | 11
Completed | 102 | 94 | 124 | 9
Not Completed | 167 | 170 | 222 | 2
Not completed — Adverse Event | 13 | 14 | 19 | 1
Not completed — Death | 1 | 1 | 3 | 0
Not completed — Lack of Efficacy | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 4 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 20 | 29 | 1
Not completed — Discontinuation of Study by Sponsor | 130 | 118 | 155 | 0
Not completed — Failed to Return | 0 | 0 | 2 | 0
Not completed — Loss of Caregiver | 0 | 1 | 3 | 0
Not completed — Vasogenic Edema Recurrence | 0 | 3 | 0 | 0
Not completed — Other | 6 | 6 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one infusion or portion of an infusion of study drug.
Groups:
- Bapineuzumab 0.5 mg/kg: Participants received 0.5 mg/kg bapineuzumab by IV infusion every 13 weeks, for a total of 6 infusions over the course of the study. A final follow-up visit was performed at Week 78, 13 weeks after the last infusion.
- Total: Total of all reporting groups
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo | Bapineuzumab 2.0 mg/kg | Total
Number analyzed (Participants) | 267 | 263 | 344 | 11 | 885
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (9.38) | 70.8 (9.73) | 69.9 (9.76) | 66.5 (7.94) | 70.6 (9.63)
Age, Customized [Number; unit: Years]
  <65 years | 73 | 81 | 115 | 6 | 275
  ≥65 years | 194 | 182 | 229 | 5 | 610
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 150 | 199 | 4 | 504
  Male | 116 | 113 | 145 | 7 | 381

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)/11 Total Score at Week 78
Description: The ADAS-Cog is a multi-item, objective measure of cognitive function. The scale evaluates memory, language, and praxis with items such as orientation, word recall, word recognition, object identification, comprehension, and the completion of simple tasks. Analysis of the ADAS-Cog for this study was based upon an 11 item score from the following items 1) word recall task, 2) naming objects and fingers, 3) following commands, 4) constructional praxis, 5) ideational praxis, 6) orientation, 7) word recognition, 8) remembering test instructions, 9) spoken language ability, 10) word finding difficulty in spontaneous speech, and 11) comprehension. This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced. The ADAS-Cog/11 ranged from 0 to 70 points, with higher scores indicating a greater degree of impairment. A negative change from baseline indicates a decrease in cognitive impairment.
Time Frame: 78 weeks
Population: The modified intent-to-treat (mITT) included all randomized participants who received at least one infusion or portion of an infusion of study drug and who had a baseline and at least one post-baseline assessment of the ADAS-Cog/11 total score and Disability Assessment for Dementia (DAD) total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Units on a scale | 6.05 (0.71) | 8.07 (0.73) | 7.88 (0.64)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Change from baseline in ADAS-Cog/11 total score was analyzed using a restricted maximum likelihood (REML) based mixed model for repeated-measures (MMRM). The number of participants in each group provided approximately 90% power to detect a 2.65 point advantage at Week 78. This calculation was based on a 2-sided test with alpha set at 0.05, the use of the Hochberg procedure to control for multiplicity; Test type: Superiority or Other; p = 0.057, Mixed Models Analysis — The p-value is not adjusted for multiple comparison. The Hochberg approach is used to control for multiplicity between the two dose levels (0.5 mg/kg and 1.0 mg/kg) of bapineuzumab; Mean Difference (Final Values) = -1.83, 95% CI 2-sided [-3.71 to 0.05]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Change from baseline in ADAS-Cog/11 total score was analyzed using a REML based MMRM. The number of participants in each group provided approximately 90% power to detect a 2.65 point advantage at Week 78. This calculation was based on a 2-sided test with alpha set at 0.05, the use of the Hochberg procedure to control for multiplicity; Test type: Superiority or Other; p = 0.848, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.73 to 2.10]

2. Primary Outcome: The Change From Baseline in the Disability Assessment for Demential (DAD) Total Score at Week 78
Description: The DAD measures instrumental and basic activities of daily living in participants with Alzheimer's Disease (AD). The DAD is administered to the participants'caregiver in the form of an interview. This scale had to be administered by a trained and certified global rater who did not have access to any information regarding adverse events experienced by the participant. This scale assesses a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item can be scored as 1 = yes, 0 = no, non applicable = NA. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores indicate better function; a positive change from baseline indicates an improvement.
Time Frame: 78 weeks
Population: The Modified Intent-to-Treat (mITT) population included as all randomized participants who received at least one infusion or portion of an infusion of study drug and who had a baseline and at least one post-baseline assessment of the ADAS-Cog/11 total score and DAD total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Units on a scale | -14.58 (1.50) | -15.07 (1.55) | -16.08 (1.36)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Change from baseline in DAD total score was analyzed using a REML based MMRM. The number of participants in each group provided approximately 90% power to detect a 6.56 point advantage at Week 78. This calculation was based on a 2-sided test with alpha set at 0.05, the use of the Hochberg procedure to control for multiplicity; Test type: Superiority or Other; p = 0.459, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [-2.48 to 5.49]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.623, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-3.04 to 5.07]

3. Secondary Outcome: The Change From Baseline in Brain Amyloid Burden at Week 71.
Description: Brain amyloid burden as imaged by 11C-Pittsburgh compound B (PiB) positron emission tomography (PET). The latter is a semiquantitative measure of the extent of fibrillar amyloid in the brain. PIB PET measurements were made in cortical regions found to have the highest burden of fibrillar amyloid at autopsy in participants diagnosed as having Alzheimer's pathology, and also regions reported to have the highest average retention of PIB signal in previous PET studies enrolling participants with probable AD. This parameter reflects overall brain amyloid deposition as indexed by imaging. The change from baseline was measured as average standard uptake value ratio (SUVr) in prespecified regions of interest (ROI) assessed by PIB PET imaging in a subset of participants.
Time Frame: 71 Weeks
Population: PiB PET population included all randomized participants who enrolled in the PET substudies and who met the following criteria: a) received at least one infusion or portion of an infusion of study drug, b) had a baseline and at least one post baseline PiB PET assessment, and c) had an SUVr for the global cortical average (GCA) ROI≥1.35 at baseline.
Measure: Least Squares Mean (Standard Error); unit: SUVr
Groups:
- Pooled Bapineuzumab 0.5/1.0 mg/kg: Participants in the bapineuzumab 0.5 and 1.0 mg/kg groups were combined to form the Pooled Bapineuzumab group.
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo | Pooled Bapineuzumab 0.5/1.0 mg/kg
Number analyzed (Participants) | 6 | 11 | 13 | 17
SUVr | -0.04 (0.08) | 0.00 (0.05) | 0.02 (0.04) | -0.01 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Pooled Bapineuzumab 0.5/1.0 mg/kg; The analysis is based on the pooled bapineuzumab (with subjects in the bapineuzumab 0.5 and 1.0 mg/kg groups combined) treatment difference estimated at Week 71. The number of participants gave 90% power to detect a 0.186 unit advantage for a bapineuzumab dose group over placebo for PiB PET binding at Week 71. The calculations were based on 2-sided tests with alpha set at 0.05 and the use of the Hochberg procedure to control for multiplicity for 2 individual doses; Test type: Superiority or Other; p = 0.654, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.15 to 0.09]

4. Secondary Outcome: The Change From Baseline in Phospho-tau Levels in the Cerebrospinal Fluid (CSF) at Week 71.
Description: Biomarkers CSF phospho-tau (p-tau) is an indicator of neuronal injury and neurodegeneration. An elevation in levels of tau, as well as specific p-tau species, is thought to be a marker for progressive cellular degeneration in AD. Accordingly, a reduction from baseline in levels of CSF tau in participants who received bapineuzumab compared with participants who received placebo may be indicative of a reduction in neuronal loss in participants treated with bapineuzumab.
Time Frame: 71 Weeks
Population: CSF population included all randomized participants who enrolled in the CSF substudies, received at least one infusion or portion of an infusion of study drug, and had a baseline and at least one postbaseline CSF measurement (CSF phospho-tau).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Groups:
- Pooled Bapineuzumab 0.5/1.0 mg/kg: Participants in the bapineuzumab 0.5 and 1.0 mg/kg groups were combined
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo | Pooled Bapineuzumab 0.5/1.0 mg/kg
Number analyzed (Participants) | 21 | 22 | 33 | 43
pg/mL | -6.62 (3.90) | -6.35 (3.73) | 0.70 (3.03) | -6.48 (2.67)
Statistical Analysis 1: Comparison: Placebo vs Pooled Bapineuzumab 0.5/1.0 mg/kg; The analysis is based on the pooled bapineuzumab (with subjects in the bapineuzumab 0.5 and 1.0 mg/kg groups combined) treatment difference estimated at Week 71. The number of participants gave 90% power to detect a 15 ng/L advantage in p-tau for a bapineuzumab dose group over placebo at Week 71. The calculations were based on 2-sided tests with alpha set at 0.05 and the use of the Hochberg procedure to control for multiplicity for 2 individual doses; Test type: Superiority or Other; p = 0.085, ANCOVA; Mean Difference (Final Values) = -7.18, 95% CI 2-sided [-15.38 to 1.02]

5. Secondary Outcome: The Change From Baseline in Brain Volume at Week 71
Description: Brain volume was examined in a subset of participants by Magnetic Resonance Imaging Brain Boundary Shift Integral (MRI BBSI). Cerebral atrophy correlates closely with the gradual cognitive decline in AD and can be visualized by MRI. The BBSI technique involves positional matching of serial 3-dimensional MRI brain images, such that brain MRI-image volumes were first registered and then subtracted from each other. Atrophy rates would generally be expected to be lower if the underlying disease was attenuated by effective treatment.
Time Frame: 71 Weeks
Population: The vMRI population Included all randomized participants who enrolled in the vMRI substudies, received at least one infusion or portion of an infusion of study drug, and had a baseline and at least one postbaseline vMRI that passed quality control and was satisfactory for volumetric analysis.
Measure: Least Squares Mean (Standard Error); unit: mL/year
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 122 | 121 | 153
mL/year | 18.55 (0.97) | 18.60 (1.00) | 17.54 (0.86)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Change in MRI BBSI was analyzed using a REML based MMRM. The number of participants gave 90% power to detect a 5.05-cm3 advantage for a bapineuzumab dose group over placebo on reduction in brain volume as measured by the BBSI at Week 71. The calculations were based on 2-sided tests with alpha set at 0.05 and the use of the Hochberg procedure to control for multiplicity for 2 individual doses; Test type: Superiority or Other; p = 0.437, Mixed Models Analysis; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-1.55 to 3.57]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.423, Mixed Models Analysis; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [-1.54 to 3.66]

6. Secondary Outcome: Divergence of Effect on the ADAS-Cog/11 Total Scores From Week 39 to Week 78
Description: The MMRM estimated slope (based on linear contrasts) of the differences between bapineuzumab and placebo for the ADAS-Cog/11 total scores from Week 39 to Week 78 was presented.
Time Frame: 39 Weeks
Population: The mITT included all randomized participants who received at least one infusion or portion of an infusion of study drug and who had a baseline and at least one post-baseline assessment of the ADAS-Cog/11 total score and DAD total score.
Measure: Mean (Standard Error); unit: Units/Year
Groups:
- Bapineuzumab 0.5 mg/kg - Placebo; Bapineuzumab 1.0 mg/kg - Placebo: For the ADAS-Cog/11 total score, results are presented from a REML based MMRM.
Arm/Group | Bapineuzumab 0.5 mg/kg - Placebo | Bapineuzumab 1.0 mg/kg - Placebo
Number analyzed (Participants) | 583 | 581
Units/Year | -1.32 (1.06) | 0.38 (1.09)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg - Placebo; Test type: Superiority or Other; p = 0.212, Mixed Models Analysis; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-3.40 to 0.76]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg - Placebo; Test type: Superiority or Other; p = 0.725, Mixed Models Analysis; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-1.76 to 2.52]

7. Secondary Outcome: Divergence of Effect on the DAD Total Scores From Week 39 to Week 78
Description: The MMRM estimated slope (based on linear contrasts)of the differences between bapineuzumab and placebo for the DAD total scores from Week 39 to Week 78 was presented.
Time Frame: 39 weeks
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Units/Years
Groups:
- Bapineuzumab 0.5 mg/kg - Placebo: For the DAD total score, results are presented from a REML-based MMRM.
- Bapineuzumab 1.0 mg/kg - Placebo: For the DAD total score, results are presented from a REML)-based MMRM.
Arm/Group | Bapineuzumab 0.5 mg/kg - Placebo | Bapineuzumab 1.0 mg/kg - Placebo
Number analyzed (Participants) | 583 | 581
Units/Years | 3.20 (2.22) | 2.01 (2.27)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg - Placebo; Test type: Superiority or Other; p = 0.149, Mixed Models Analysis; Mean Difference (Final Values) = 3.20, 95% CI 2-sided [-1.15 to 7.56]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg - Placebo; Test type: Superiority or Other; p = 0.375, Mixed Models Analysis; Mean Difference (Final Values) = 2.01, 95% CI 2-sided [-2.44 to 6.46]

8. Secondary Outcome: Time to Median Placebo Deterioration on ADAS-Cog/11 Total Score (European Union [EU] Analysis Plan)
Description: The time to first median placebo deterioration (for the EU) was defined as the first time a subject experienced an increase from baseline (worsening) in ADAS Cog/11 total score greater than or equal to the median worsening observed at Week 78 in the placebo group. The Kaplan Meier estimate of the median time to first median placebo deterioration in ADAS Cog/11 total score was presented.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Days | 546.0 [546.0 to NA] — Value was not calculable due to the large number of censored event times | 462.0 [455.0 to 546.0] | 540.0 [462.0 to 546.0]
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.030, Log Rank — Not specifed
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.567, Log Rank

9. Secondary Outcome: Time to First Clinically Meaningful Deterioration on ADAS-Cog/11 Total Score (United States [US] Analysis Plan)
Description: The time to first clinically meaningful deterioration (for the US) was defined as the first time a participant experienced an increase (worsening) from baseline in ADAS-Cog/11 total score of >=7.
Time Frame: 78 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Days | 546.0 [546.0 to NA] — Values were not calculable due to the large number of censored event times | 546.0 [455.0 to 546.0] | 546.0 [476.0 to 546.0]
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.079, Log Rank
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.675, Log Rank

10. Secondary Outcome: Time to Median Placebo Deterioration on DAD Total Score
Description: The time to first median placebo deterioration (for the EU) was defined as the first time a participant experienced a decrease (worsening) in DAD total score greater than or equal to the median worsening at Week 78 in the placebo group.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Days | 541.0 [455.0 to 546.0] | 534.0 [372.0 to NA] — Values were not calculable due to the large number of censored event times | 463.0 [453.0 to 546.0]
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Not spsecified; Test type: Superiority or Other; p = 0.846, Log Rank
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.797, Log Rank

11. Secondary Outcome: Time to First Clinically Meaningful Deterioration on DAD Total Score (US Analysis Plan)
Description: The time to first clinically meaningful deterioration was defined as the first time a participant experienced a decrease (worsening)from baseline in DAD total score of >=12.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Days | 542.0 [456.0 to 546.0] | 539.0 [450.0 to NA] — Value was not calculable due to the large number of censored event times | 540.0 [453.0 to 546.0]
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.933, Log Rank
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.714, Log Rank

12. Secondary Outcome: Percentage of Participants With Worsening From Baseline in ADAS-Cog/11 Total Score at Week 78 (European Union Analysis Plan)
Description: Percentage of participants whose increase (worsening) in ADAS-Cog/11 total score from baseline to Week 78 was at most 0, 3, 7 points.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Number of participants
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Number of participants
  Worsening of 0 points | 10.6 [7.1 to 15.0] | 8.7 [5.5 to 12.9] | 7.3 [4.7 to 10.7]
  Worsening of 3 points | 16.1 [11.8 to 21.2] | 13.4 [9.5 to 18.3] | 10.1 [7.0 to 13.8]
  Worsening of 7 points | 23.1 [18.1 to 28.8] | 19.0 [14.3 to 24.4] | 19.2 [15.1 to 23.9]

13. Secondary Outcome: Percentage of Participants With Worsening From Baseline in ADAS-Cog/11 Total Score at Week 78 (US Analysis Plan)
Description: Percentage of participants whose increase (worsening) from baseline to Week 78 in ADAS-Cog/11 total score is <7.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Percentage of participants | 22.4 | 18.6 | 18.6
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.277, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.996, Cochran-Mantel-Haenszel

14. Secondary Outcome: Percentage of Participants With Worsening From Baseline in DAD Total Score at Week 78 (European Union Analysis Plan)
Description: Percentage of participants whose decrease (worsening) from baseline to Week 78 in DAD total score was at most 0, 6, 12 points.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Percentage of participants
  Worsening of 0 points | 10.2 [6.8 to 14.6] | 11.9 [8.1 to 16.5] | 9.1 [6.3 to 12.8]
  Worsening of 6 points | 15.7 [11.4 to 20.7] | 16.6 [12.2 to 21.8] | 14.3 [10.7 to 18.6]
  Worsening of 12 points | 20.0 [15.3 to 25.4] | 22.1 [17.2 to 27.8] | 19.5 [15.4 to 24.2]

15. Secondary Outcome: Percentage of Participants With Worsening From Baseline in DAD Total Score at Week 78 (US Analysis Plan)
Description: Percentage of participants whose decrease (worsening) from baseline to Week 78 in DAD total score was <12.
Time Frame: 78 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Percentage of participants | 20.0 | 22.1 | 19.5
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.855, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.423, Cochran-Mantel-Haenszel

16. Secondary Outcome: Change From Baseline in Dependence Scale Total Score at Week 78
Description: The Dependence Scale (DS) is a 13-item, caregiver-rated instrument for determining the amount of support required by a participant with AD. The DS total score ranges from 0 to 15, with higher scores indicating more need for assistance. The DS was administered as an interview to the caregiver at scheduled study visits.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Units on a scale | 1.29 (0.19) | 1.16 (0.19) | 1.45 (0.17)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Change in DS score was analyzed using a REML based MMRM; Test type: Superiority or Other; p = 0.516, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.65 to 0.33]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Change in DS score was analyzed using a REML based MMRM; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.79 to 0.21]

17. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SOB) Total Score at Week 78
Description: The CDR-SOB is a global clinical staging instrument that sums 6 clinical ratings: 1) memory, 2) orientation, 3) judgment and problem solving, 4) involvement in community affairs, 5) home and hobbies, and 6) personal care based on the Clinical Dementia Rating Scale (CDR) interview. The CDR includes discussions with the participant and caregiver using a structured format. This scale had to be administered by a trained and certified global rater who did not have access to any information regarding adverse events experienced by the participant. CDR-SOB total score range is 0 (least impairment) to 18 (most impairment); a negative change from baseline indicates an improvement.
Time Frame: 78 Weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo
Number analyzed (Participants) | 255 | 253 | 328
Units on a scale | 2.23 (0.23) | 2.41 (0.23) | 2.59 (0.20)
Statistical Analysis 1: Comparison: Bapineuzumab 0.5 mg/kg vs Placebo; Change in CDR-SOB total score was analyzed using a REML based MMRM; Test type: Superiority or Other; p = 0.238, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.96 to 0.24]
Statistical Analysis 2: Comparison: Bapineuzumab 1.0 mg/kg vs Placebo; Change in CDR-SOB total score was analyzed using a REML based MMRM; Test type: Superiority or Other; p = 0.564, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.78 to 0.43]

ADVERSE EVENTS:
Time Frame: 4 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Bapineuzumab 2.0 mg/kg: Participants received placebo by IV infusion every 13 weeks, for a total of 6 infusions over the course of the study. A final follow-up visit was performed at Week 78, 13 weeks after the last infusion.
Arm/Group | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Placebo | Bapineuzumab 2.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 32/267 | 34/263 | 53/344 | 2/11
Other Adverse Events (participants affected / at risk) | 109/267 | 123/263 | 124/344 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bapineuzumab 0.5 mg/kg (N=267) | Bapineuzumab 1.0 mg/kg (N=263) | Placebo (N=344) | Bapineuzumab 2.0 mg/kg (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adams-Stokes syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heat illness (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECG signs of myocardial ischaemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Perineurial cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural hygroma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 6 (8) | 12 (20) | 0 (0) | 2 (7)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jealous delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bapineuzumab 0.5 mg/kg (N=267) | Bapineuzumab 1.0 mg/kg (N=263) | Placebo (N=344) | Bapineuzumab 2.0 mg/kg (N=11)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (4) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (16) | 6 (6) | 9 (10) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 7 (7) | 11 (15) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (11) | 9 (11) | 10 (12) | 3 (3)
Catheter site haematoma (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 17 (23) | 18 (24) | 28 (44) | 2 (2)
Sinusitis (Infections and infestations) | 5 (16) | 3 (3) | 3 (5) | 1 (12)
Urinary tract infection (Infections and infestations) | 15 (17) | 13 (17) | 9 (13) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 8 (10) | 1 (1) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 18 (25) | 16 (18) | 18 (26) | 1 (1)
Blood pressure increased (Investigations) | 5 (5) | 5 (9) | 6 (7) | 2 (3)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (15) | 5 (17) | 6 (9) | 1 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 2 (4) | 2 (6) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral microhaemorrhage (Nervous system disorders) | 11 (13) | 22 (41) | 9 (21) | 1 (9)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 7 (20) | 16 (17) | 1 (5)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Exertional headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 17 (19) | 15 (36) | 29 (36) | 2 (9)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Vasogenic cerebral oedema (Nervous system disorders) | 7 (16) | 20 (43) | 2 (7) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 3 (5) | 6 (6) | 1 (3)
Depression (Psychiatric disorders) | 13 (25) | 11 (21) | 9 (24) | 2 (9)
Hallucination (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 10 (12) | 9 (16) | 2 (9)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The impact of study termination, the shorter observational periods and the resulting small sample size coupled with not having enough participants with post baseline assessments for various reasons were limiting factors for data interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.